CLINICAL TRIAL: NCT04838951
Title: Effect of Real-time Computer-aided System (ENDO-AID) on Adenoma Detection in Endoscopist-in-training: a Single-blind Randomized Study
Brief Title: Effect of Real-time Computer-aided System (ENDO-AID) on Adenoma Detection in Endoscopist-in-training
Acronym: ENDOAIDTRAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Louis Ho Shing Lau, Resident Specialist, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021.141
Record Dates: First submitted 2021-03-23; First posted 2021-04-09 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Screening Colonoscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Endoscopist wil not be blinded to treatment. Treatment arm allocation will be concealed to patients, data collector and data analysts.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): CADe system will be used during withdrawal phase of colonoscopy.
  Interventions: Device: ENDO-AID CADe
- Control arm (No Intervention): Colonoscopy will be performed according to hospital protocol.

INTERVENTIONS:
Device: ENDO-AID CADe — ENDO-AID CADe will be used during the withdrawal process of the colonoscopy.
  Arms: Intervention arm

SUMMARY:
The investigator's hypothesis is that a CADe system (ENDO-AID) would improve the adenoma detection rate in junior endoscopists.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the most common and second most lethal cancer in Hong Kong with more than 5,600 new cases and 2,300 deaths annually. Colonoscopy with polypectomy has shown to reduce CRC-related mortality by 53%. However, high polyp miss rates were reported to be up to 26% for adenomas and 9% for advanced adenomas in standard colonoscopies. Risk factors included proximal location, serrate or flat lesions, poor bowel preparation and short withdrawal time (<6 minutes). Insufficient trainee experience was also associated with a higher adenoma miss rate. A significant proportion of interval CRC was attributed to the missed lesions during index colonoscopy leading to adverse patient outcomes.

As a result, various techniques were developed to improve adenoma detection rate (ADR) during colonoscopies. Techniques including water exchange method, second examination of the right colon (retroflexion or second forward view)and cap/cuff-assisted colonoscopies were proven to increase ADR effectively. However, these techniques were operator-dependent requiring certain level of expertise.

Recently, artificial intelligence and computer-aided polyp detection (CADe) systems have developed rapidly around the globe. These systems can provide real-time CADe by flagging the suspected lesions to endoscopists, with the adoption of deep learning or convoluted neural networks. A number of prospective randomized clinical trials reported a significant increase in ADR in CADe group. The number of adenoma detected per colonoscopy was consistently higher among different polyp sizes, location and morphology. The ADR increment was particularly higher for diminutive adenomas smaller than 5mm.

Nevertheless, most of the aforementioned studies only involved senior endoscopists for the procedures. Theoretically, the senior endoscopists were more skillful to expose colonic mucosa and more experienced to distinguish the false positive computer signals, leading to an enhanced performance of CADe in real-time colonoscopies. The effect of CADe on inexperienced junior endoscopists performing colonoscopies remains largely unknown.

In this single-blind randomized study, the investigators aim to evaluate the effect of a new CADe system (ENDO-AID) on adenoma detection and quality improvement in junior endoscopists.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years old or above;
2. They require elective colonoscopy for colorectal cancer screening, polyp surveillance, or investigation of symptoms such as anemia or gastrointestinal bleeding;
3. Written informed consent obtained.

Exclusion Criteria:

1. Contraindication to colonoscopy (e.g. intestinal obstruction or perforation)
2. Contraindication or conditions precluding polyp resection (e.g. active gastrointestinal bleeding, significant bleeding tendency, uninterrupted anticoagulation or dual antiplatelets)
3. Scheduled staged procedure for polypectomy or biopsy
4. Previous colonic resection
5. Personal history of colorectal cancer
6. Personal history of polyposis syndrome
7. Personal history of inflammatory bowel disease
8. Advanced comorbid conditions (defined as American Society of Anesthesiologists grade 4 or above)
9. Pregnancy
10. Unable to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 856 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-07-22 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
ADR | During the colonoscopy
  adenoma detection rate

SECONDARY OUTCOMES:
ADR for adenomas of different sizes | During the colonoscopy
  <5mm, 5-10mm, >10mm
ADR for adenomas of different colonic segments | During the colonoscopy
  caecum, ascending colon, hepatic flexure, transverse colon, splenic flexure, descending colon, sigmoid colon, rectum
Mean number of adenomas per colonoscopy | During the colonoscopy
  Mean number of adenomas per colonoscopy
Advanced adenoma detection rate | During the colonoscopy
  Advanced adenoma detection rate
Sessile serrate lesion (SSL) detection rate | During the colonoscopy
  Sessile serrate lesion (SSL) detection rate
Polyp detection rate | During the colonoscopy
  Polyp detection rate
Non-neoplastic resection rate | During the colonoscopy
  defined as absence of adenoma or SSL within resected specimen
Missed polyp rate | During the colonoscopy
  defined as a polyp which the junior endoscopist fails to recognize and withdraws the endoscope to next colonic segment, but detected by the supervisor
False positive rate | During the colonoscopy
  defined as computer artifacts due to colonic mucosal wall or bowel content lasting for >2 seconds
Cecal intubation time | During the colonoscopy
  Cecal intubation time
Withdrawal time | During the colonoscopy
  excluding interventions
Total procedural time | During the colonoscopy
  Total procedural time
Percentage of change in ADR in relation to the personal experience in colonoscopy | During the colonoscopy
  Percentage of change in ADR in relation to the personal experience in colonoscopy based on number of procedures performed <200 vs 200-500

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, New Territories, Hong Kong

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data to other researchers

REFERENCES:
- [Derived] Lau LHS, Ho JCL, Lai JCT, Ho AHY, Wu CWK, Lo VWH, Lai CMS, Scheppach MW, Sia F, Ho KHK, Xiao X, Yip TCF, Lam TYT, Kwok HYH, Chan HCH, Lui RN, Chan TT, Wong MTL, Ho MF, Ko RCW, Hon SF, Chu S, Futaba K, Ng SSM, Yip HC, Tang RSY, Wong VWS, Chan FKL, Chiu PWY; ENDOAID-TRAIN study group. Effect of Real-Time Computer-Aided Polyp Detection System (ENDO-AID) on Adenoma Detection in Endoscopists-in-Training: A Randomized Trial. Clin Gastroenterol Hepatol. 2024 Mar;22(3):630-641.e4. doi: 10.1016/j.cgh.2023.10.019. Epub 2023 Nov 2. PMID 37918685